CLINICAL TRIAL: NCT06504875
Title: Application of PD-1 Monoclonal Antibody in Combination With IL-2 and CapeOX in Organ Preservation Therapy for Ultra-Low Localized Advanced Rectal Cancer: A Single-center, Single-arm, Open-label Clinical Study (PICTURE)
Brief Title: Application of PD-1 Monoclonal Antibody in Combination With IL-2 and CapeOX in Organ Preservation Therapy for Ultra-Low Localized Advanced Rectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: PICTURE202407
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Rectal Cancer
Keywords: Tislelizumab; Interleukin-2; MSS/pMMR rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — tislelizumab; Interleukin-2; Capecitabine; Oxaliplatin

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CapeOX+PD-1+IL-2: Tislelizumab 200mg ivd D1 + Interleukin 2 100IU HD,QOD d1-d14 +CapeOX (Capecitabine: 1000mg/m2 bid po, d1-d14；Oxaliplatin 130mg/m2 ivd, d1) 6 cycles
  Interventions: Drug: Tislelizumab; Drug: Interleukin-2; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg ivd D1
Drug: Interleukin-2 — Interleukin 2 100IU HD,QOD d1-d14
Drug: Capecitabine — Capecitabine: 1000mg/m2 bid po, d1-d14
Drug: Oxaliplatin — Oxaliplatin 130mg/m2 ivd, d1

SUMMARY:
The objective is to evaluate whether the neoadjuvant combination of PD-1 inhibitor tislelizumab and interleukin-2 (IL-2) can significantly enhance the complete response rate (cCR + local excision pCR) and organ preservation rate in patients with MSS/pMMR locally advanced rectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) stands as a prominent global health concern, ranking among the most prevalent malignancies worldwide. Its incidence exhibits striking geographical variations, with higher rates observed in developed countries. Age is a significant risk factor, predominantly affecting individuals aged 50 and above, although a concerning trend of increasing incidence in younger adults has been noted in recent years. There exists a gender disparity, with slightly higher prevalence in males. Notably, lifestyle factors, including dietary choices, sedentary habits, smoking, and obesity, play crucial roles in its etiology. These epidemiological patterns underscore the urgency for implementing effective prevention strategies and advancing early detection methods to mitigate the disease's impact.

In China, nearly two-thirds of colorectal cancer cases are rectal cancers, with approximately half being low rectal cancers. Currently, surgical resection remains the primary curative approach for patients with low rectal cancer. The concept of Total Mesorectal Excision (TME), introduced in 1982, has become the standard surgical procedure for low rectal cancer, focusing on en bloc removal of the rectum along with its mesentery to reduce the local recurrence rate post-surgery. Building upon this, the advent of neoadjuvant chemoradiotherapy, watch-and-wait strategies, targeted therapies, and immunotherapies has shifted the focus of low rectal cancer management from merely increasing R0 resection rates and decreasing local tumor recurrence to encompassing precise imaging-based staging, efficacy assessment, organ function preservation, and quality-of-life improvements.

In colorectal cancer, the PD-1 inhibition pathway plays a central role in regulating immune cell exhaustion. However, monotherapy targeting PD-1 alone shows limited responses in most colorectal cancer patients, suggesting that combinations with other immunostimulatory agents could address this challenge. Several combinatorial approaches have shown promise in animal models and are now being explored in clinical settings. Among these, Interleukin-2 (IL-2) is emerging as a potential candidate to synergize with PD-1 blockade in exerting antitumor effects. Our study aims to explore the synergy of IL-2 combined with a PD-1 inhibitor, seeking to overcome the limitations of single-agent immunotherapy through multifaceted immune modulation. By enhancing immune cell infiltration and disrupting the physical and immunosuppressive barriers of tumors, we aim to augment the efficacy of immunotherapy and increase the organ preservation rate in ultra-low locally advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤75 years
2. Histologically confirmed adenocarcinoma of the rectum
3. pMMR (proficient mismatch repair) or MSI-L (microsatellite instability-low) or MSS (microsatellite stable)
4. Tumor distance from the anal verge ≤5 cm
5. Clinical stage of cT1-3N1M0 or cT2-3N0M0
6. ECOG performance status score ≤ 1

Exclusion Criteria:

1. Patients with metastatic disease (Stage IV); recurrent colorectal cancer with active bleeding, perforation, or complex conditions requiring urgent surgery; or concurrent non-colorectal cancer malignancies.
2. Patients who have previously received systemic anticancer therapy for colorectal cancer; or have been treated with PD-1, PD-L1, or CTLA-4 antibodies.
3. Patients with any active autoimmune disease; known or tested positive for Human Immunodeficiency Virus (HIV) or Acquired Immunodeficiency Syndrome (AIDS); or a history requiring steroid or immunosuppressive drug treatment.
4. Patients with interstitial lung disease, non-infectious pneumonitis, or uncontrolled systemic diseases (such as diabetes, hypertension, pulmonary fibrosis, and acute pneumonia).
5. Patients who experienced any Grade 2 or higher toxicities due to prior treatments (as classified by the Common Terminology Criteria for Adverse Events [CTCAE] version 5), which have not resolved (excluding anemia, alopecia, and skin pigmentation changes); known or suspected history of hypersensitivity to any of the drugs used in the trial.
6. Pregnant or breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Age ≥18 years and ≤75 years
  2. Histologically confirmed adenocarcinoma of the rectum
  3. pMMR (proficient mismatch repair) or MSI-L (microsatellite instability-low) or MSS (microsatellite stable)
  4. Tumor distance from the anal verge ≤5 cm
  5. Clinical stage of cT1-3N1M0 or cT2-3N0M0
  6. ECOG performance status score ≤ 1
Sampling Method: Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2024-07-10 (Estimated); Primary Completion 2025-07-10 (Estimated); Study Completion 2027-07-10 (Estimated)

PRIMARY OUTCOMES:
CR rate (cCR + local excision pCR) | 1 years
  Complete Response rate," which includes both "complete clinical response" (cCR) and "pathologic complete response after local excision" (pCR)

SECONDARY OUTCOMES:
organ preservation rates | 1 month
  The assessment of how different treatment strategies, determined by the Complete Response (CR) status post-neoadjuvant chemotherapy, affect the anal sphincter preservation in patients with locally advanced low rectal cancer.
Event-Free Survival rates | 5 years
  Event-Free Survival (EFS) is the length of time after treatment during which the patient survives without any events of interest occurring, such as disease progression, recurrence, or death. Therefore, the 1/2/3-year EFS rates refer to the percentages of patients surviving without these events at 1, 2, and 3 years.
Overall Survival rates | 5 year
  Overall Survival (OS) is the most common endpoint in cancer clinical trials, measuring the proportion of patients still alive at specific time points after the start of treatment. Thus, the 1/2/3-year OS rates represent the percentages of patients still alive at 1, 2, and 3 years post-treatment.

IPD SHARING:
Plan to Share IPD: Undecided